CLINICAL TRIAL: NCT04316117
Title: FDG PET to Assess Therapeutic Response in Patients With Bone-Dominant Metastatic Breast Cancer, FEATURE
Brief Title: Using FDG-PET/CT to Assess Response of Bone-Dominant Metastatic Breast Cancer, FEATURE Study
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EA1183; NCI-2020-00210 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA1183 (Other: ECOG-ACRIN Cancer Research Group); EA1183 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Hormone Receptor Positive Breast Carcinoma; Metastatic Breast Carcinoma; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Systemic therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (FDG-PET/CT) (Experimental): Patients receive FDG IV and undergo PET/CT scan over 15-30 minutes at baseline (within 21 days before start of standard systemic treatment) and at 12 weeks after start of standard systemic treatment in the absence of unacceptable toxicity.
  Interventions: Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT scan; computerized axial tomography; Computerized Tomography; CT; CT scan; tomography
Other: Fludeoxyglucose F-18 — Given IV
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; positron emission tomography scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well FDG-PET/CT works in assessing the response of patients with breast cancer that has spread to the bones or mostly to the bones (bone-dominant metastatic breast cancer). Diagnostic procedures, such as FDG-PET/CT, may work better in measuring breast cancer activity before and after treatment compared to other standard imaging tests.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Evaluate the performance of fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) response criteria (modified PET Response Criteria in Solid Tumors [PERCIST] complete, partial and stable metabolic disease versus progressive metabolic disease) as a binary predictor of progression-free survival (PFS) in patients with bone-dominant (BD) metastatic breast cancer (MBC) treated with systemic therapy.

SECONDARY OBJECTIVES:

I. Evaluate the ability of FDG-PET/CT modified PERCIST criteria (complete versus [vs] partial vs stable vs metabolic progression) to independently predict PFS in patients with BD MBC.

II. Evaluate the ability of FDG-PET/CT modified PERCIST criteria (complete, partial, and stable versus progressive metabolic disease) to predict time to skeletal related events (SRE) and overall survival (OS) in patients with BD MBC.

III. Evaluate the ability of FDG-PET/CT metrics (percent change in peak standardized uptake value corrected for lean body mass (SULpeak), maximum standardized uptake value corrected for body weight (SUVmax) as continuous variables in index or up to 5 lesions) to predict PFS, time to SRE and OS in patients with BD MBC.

IV. Assess the utility of FDG-PET/CT to identify disease progression by identification of new lesions not identified by standard CT and bone scan.

EXPLORATORY OBJECTIVES:

I. Define criteria for selection of FDG-avid bone lesions for analysis based on thresholds for SULpeak or SUVmax.

II. In collaboration with National Cancer Institute (NCI) Quantitative Imaging Network (QIN), explore alternative methods for measuring metabolic response with FDG-PET/CT (e.g., total lesion glycolysis, quantitative total bone imaging, MD Anderson bone criteria, and radiomics) to predict clinical endpoints in patients with BD MBC.

III. Evaluate automated image analysis of FDG-PET/CT by AutoPERCIST.

OUTLINE:

Patients receive FDG intravenously (IV) and undergo PET/CT scan over 15-30 minutes at baseline (within 21 days before start of standard systemic treatment) and at 12 weeks after start of standard systemic treatment in the absence of unacceptable toxicity.

After completion of study, patients are followed up periodically for up to 3 years after study registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance (performance status [PS]) =< 2
* Patients with histologically confirmed metastatic breast cancer by local assessment that is hormone receptor positive by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines and with known HER2 status
* Patients must have radiologically confirmed bone-dominant (BD) or bone-only (BO) disease

  * BD defined as disease involving bone with or without limited measurable metastases by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, with >= 1 non-irradiated bone metastasis on bone scintigraphy

    * NOTE: Limited measurable metastases includes lymph nodes and the soft tissue components of lytic or mixed lytic/blastic bone metastases. Any number of lymph nodes < 3 cm and up to 2 lymph nodes > 3 cm will be allowed. Up to 5 measurable soft tissue components of lytic or mixed mytic/blastic bone metastases will be allowed
  * BO defined as detectable disease confined within the bone (any site, any number of lesions). Diagnosis requires abnormalities identified by imaging (bone scan, CT +/- PET +/- magnetic resonance imaging [MRI]) with no other sites of metastases identified and with >= 1 non-irradiated bone metastasis on bone scintigraphy
* Patients must have no contraindication to FDG-PET imaging
* Patients must have one of the following systemic therapies:

  * Plan to receive either 1st or 2nd line endocrine therapy for metastatic breast cancer. Endocrine therapy may include selective estrogen receptor modulators (SERMs), aromatase inhibitors, and/or fulvestrant that may be combined with Food and Drug Administration (FDA)-approved biologic agents (palbociclib, ribociclib, abemaciclib, everolimus, alpelisib)
  * Chemotherapy per National Comprehensive Cancer Network (NCCN) or institutional standard. Use of colony stimulating growth factor must be suspended for >= 14 days prior to FDG-PET/CT scans at baseline and 12-weeks
  * Plan to receive HER2-targeted therapy per ASCO, NCCN, and/or institutional guidelines as indicated for patients with HER2 positive disease. When HER2-targeted therapy is used with chemotherapy, use of colony stimulating growth factors is NOT expected or should be suspended for a minimum of 2 weeks, but preferably for at least 3 weeks prior to the required FDG-PET/CT scan time points
* The use of bone-stabilizing agents (bisphosphonates or denosumab) is permitted
* Patient must meet institutional guidelines for renal function for MRI and CT scanning
* Patient's life expectancy must be estimated at >= 24 weeks
* The patient is participating in the trial at an institution which has agreed to perform the imaging research studies, completed the ECOG-American College of Radiology Imaging Network (ACRIN) defined PET/CT scanner qualification procedures and received ECOG-ACRIN PET/CT scanner approval
* Patients must complete the baseline (T0) FDG-PET within 28 days prior to registration or within 28 days after registration

  * For patients completing the baseline (T0) FDG-PET AFTER registration all parameters must be met
  * For patients who completed the baseline (T0) FDG-PET prior to registration the following tests are exempt:

    * Pregnancy testing documentation prior to FDG-PET (T0 time point)

Exclusion Criteria:

* Patients with RECIST 1.1 measurable lesions in viscera, active central nervous system (CNS), leptomeningeal carcinomatous or pleural or peritoneal disease will not be eligible. Patients with prior CNS metastases treated with radiation or resection and without evidence of clinical or radiographic progression within 28 days of registration are eligible
* Patients who have received greater than 3 lines of cytotoxic chemotherapy for metastatic breast cancer are not eligible
* Patients currently participating in or have participated in a study of an investigational agent or using an investigational device within 3 weeks of study registration are not eligible
* Patients with known additional malignancy that is progressing or requires active treatment are not eligible. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Women must not be pregnant because FDG is a radiopharmaceutical with the potential for teratogenic effects and PET/CT involves additional radiation exposure. In addition, because of radiation exposure to a nursing infant from FDG, women who are breastfeeding are also excluded from this study. All females of childbearing potential must have a blood test or urine study within 7 days prior to FDG-PET/CT to rule out pregnancy. Patients are excluded from this if baseline FDG-PET/CT scan met study parameters and was completed within 28 days of study registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Performance of fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) response criteria as a binary predictor of progression-free survival (PFS) | Up to 3 years after study registration
  Will evaluate the performance of FDG-PET/CT response criteria (modified PET Response Criteria in Solid Tumors complete, partial and stable metabolic disease versus progressive metabolic disease) as a binary predictor of PFS in patients with bone-dominant (BD) metastatic breast cancer (MBC) treated with systemic therapy.

SECONDARY OUTCOMES:
Ability of FDG-PET/CT modified PERCIST criteria (complete versus [vs] partial vs stable vs metabolic progression) to independently predict PFS in patients with BD MBC | Up to 3 years after study registration
  Will keep the multiple categories of FDG-PET/CT modified PERCIST criteria and test the PFS differences across them using the Kaplan-Meier survival curve and the corresponding log-rank test. The multivariable Cox proportional hazard model will be also fitted with the adjustment of the same set of confounders (e.g., age, line of therapy - early line treatment versus late line treatment, type of therapy - endocrine therapy versus chemotherapy). Since the categories of FDG-PET/CT modified PERCIST criteria are ordered, will also apply the method of C-statistics to evaluate the performance after quantifying the criteria (i.e., 1-complete response, 2-partial response, 3-stable, 4-metabolic progression).
Ability of FDG-PET/CT modified PERCIST criteria (complete, partial, and stable vs progressive metabolic disease) to predict time to skeletal related events (SRE) in patients with BD MBC | Up to 3 years after study registration
  Will keep the multiple categories of FDG-PET/CT modified PERCIST criteria and test the time to SRE differences across them using the Kaplan-Meier survival curve and the corresponding log-rank test. The multivariable Cox proportional hazard model will be also fitted with the adjustment of the same set of confounders (e.g., age, line of therapy - early line treatment versus late line treatment, type of therapy - endocrine therapy versus chemotherapy). Since the categories of FDG-PET/CT modified PERCIST criteria are ordered, will also apply the method of C-statistics to evaluate the performance after quantifying the criteria (i.e., 1-complete response, 2-partial response, 3-stable, 4-metabolic progression).
Ability of FDG-PET/CT modified PERCIST criteria (complete, partial, and stable vs progressive metabolic disease) to predict overall survival (OS) in patients with BD MBC | Up to 3 years after study registration
  Will keep the multiple categories of FDG-PET/CT modified PERCIST criteria and test the OS differences across them using the Kaplan-Meier survival curve and the corresponding log-rank test. The multivariable Cox proportional hazard model will be also fitted with the adjustment of the same set of confounders (e.g., age, line of therapy - early line treatment versus late line treatment, type of therapy - endocrine therapy versus chemotherapy). Since the categories of FDG-PET/CT modified PERCIST criteria are ordered, will also apply the method of C-statistics to evaluate the performance after quantifying the criteria (i.e., 1-complete response, 2-partial response, 3-stable, 4-metabolic progression).
Ability of FDG-PET/CT metrics to predict PFS in patients with BD MBC | Up to 3 years after study registration
  For each participant, will collect up to 5 lesions from FDG-PET/CT scans and calculate the percent change in peak standardized uptake value corrected for lean body mass (SULpeak), maximum standardized uptake value corrected for body weight (SUVmax) from T0 to T1 scans. Multivariable Cox proportional hazard models will be used to model the ability of these changes to predict PFS. The analysis will first be conducted on the index lesion (i.e., associating the change of SUVpeak or SUVmax for the index lesion with outcomes), and then be applied to the average change of up to 5 lesions (i.e., associating the average change of SUVpeak or SUVmax from all detected lesions with outcomes). The C-statistics will be used to measure the performance.
Ability of FDG-PET/CT metrics to predict time to SRE in patients with BD MBC | Up to 3 years after study registration
  For each participant, will collect up to 5 lesions from FDG-PET/CT scans and calculate the percent change in SULpeak, SUVmax from T0 to T1 scans. Multivariable Cox proportional hazard models will be used to model the ability of these changes to predict time to SRE. The analysis will first be conducted on the index lesion (i.e., associating the change of SUVpeak or SUVmax for the index lesion with outcomes), and then be applied to the average change of up to 5 lesions (i.e., associating the average change of SUVpeak or SUVmax from all detected lesions with outcomes). The C-statistics will be used to measure the performance.
Ability of FDG-PET/CT metrics to predict OS in patients with BD MBC | Up to 3 years after study registration
  For each participant, will collect up to 5 lesions from FDG-PET/CT scans and calculate the percent change in SULpeak, SUVmax from T0 to T1 scans. Multivariable Cox proportional hazard models will be used to model the ability of these changes to predict OS. The analysis will first be conducted on the index lesion (i.e., associating the change of SUVpeak or SUVmax for the index lesion with outcomes), and then be applied to the average change of up to 5 lesions (i.e., associating the average change of SUVpeak or SUVmax from all detected lesions with outcomes). The C-statistics will be used to measure the performance.
Utility of FDG-PET/CT to identify disease progression by identification of new lesions not identified by standard CT and bone scan | Up to 3 years after study registration
  For the cases where progression is documented in the study, will record and tabulate the number of new lesions uniquely identified by the 12-week FDG-PET/CT research scan.

OTHER OUTCOMES:
Defining of criteria for selection of FDG-avid bone lesions for analysis based on thresholds for SULpeak or SUVmax | Up to 3 years after study registration
  Will vary the threshold for inclusion in the PERCIST criteria to get optimum performance. To reduce the over-optimism, will apply the statistical technique of 5-fold cross-validation in the threshold discovery and subsequent performance assessment.
Exploration of alternative methods for measuring metabolic response with FDG-PET/CT to predict clinical endpoints in patients with BD MBC | Up to 3 years after study registration
  Will collaborate with National Cancer Institute Quantitative Imaging Network to explore alternative methods for measuring metabolic response with FDG-PET/CT scans. Will then implement Kaplan Meier survival curve (and log-rank test) or multivariable Cox proportional hazard model in the analyses of associations with PFS, time to SRE, or OS.
Automated image analysis of FDG-PET/CT | Up to 3 years after study registration
  Will evaluate automated image analysis of FDG-PET/CT by AutoPERCIST.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Specht, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (104):
- United States (98):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - GenesisCare USA - Aventura FP, Aventura, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Jewish Hospital, Louisville, Kentucky
  - UPMC Western Maryland, Cumberland, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Cork University Hospital, Cork, Ireland
- Puerto Rico (5):
  - Cancer Center-Metro Medical Center Bayamon, Bayamón
  - Doctors Cancer Center, Manatí
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Makhlin I, Korhonen KE, Martin ML, Gillman J, Schubert E, Pantel AR, Mankoff DA, Clark AS. 18F-FDG PET/CT for the Evaluation of Therapy Response in Hormone Receptor-Positive Bone-Dominant Metastatic Breast Cancer. Radiol Imaging Cancer. 2022 Nov;4(6):e220032. doi: 10.1148/rycan.220032. PMID 36269154